CLINICAL TRIAL: NCT00002964
Title: Pilot Study for the Diagnosis of Head and Neck Cancer: Photofrin and Visible Light
Brief Title: Porfimer Sodium in Diagnosing Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Purpose: Diagnostic
Other Study IDs: DS 94-10; RPCI-DS-94-10; NCI-V97-1196
Record Dates: First submitted 1999-11-01; First posted 2004-04-27 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Head and Neck Cancer
Keywords: stage 0 oropharyngeal cancer; stage 0 laryngeal cancer; stage 0 hypopharyngeal cancer; stage 0 lip and oral cavity cancer; stage I lip and oral cavity cancer; stage I hypopharyngeal cancer; stage I laryngeal cancer; stage I oropharyngeal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms; Laryngeal Neoplasms; Hypopharyngeal Neoplasms; Mouth Neoplasms | interventions — Dihematoporphyrin Ether; Fluorophotometry

INTERVENTIONS:
Drug: porfimer sodium
Other: fluorophotometry

SUMMARY:
RATIONALE: Drugs that make cancer cells more visible to light may help in the diagnosis of head and neck cancer.

PURPOSE: Phase II trial to study the usefulness of porfimer sodium in diagnosing patients with head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether porfimer sodium fluorescence can be used to reveal early malignant changes in patients with lesions of the oral cavity. II. Investigate whether porfimer sodium fluorescence can define areas of field cancerization in the oral mucosa, specifically satellite foci of malignant cells within the margins of an excision. III. Determine whether uptake of fluorescence is indicative of disease stage.

OUTLINE: Patients receive porfimer sodium IV bolus and are kept in subdued light until examination with a fluorescence photometer 48 hours later. Patients must avoid sunlight and other intense lights for an additional 30 days.

PROJECTED ACCRUAL: 20 patients will be accrued per year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Malignant or suspected lesions of the head and neck that are scheduled for excisional biopsy Lesions no greater than 2 cm in diameter in the mouth, oropharynx, hypopharynx or larynx Suspected severe dysplasia, carcinoma in situ and/or invasive carcinoma of the head and neck

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: WBC greater than 3500/mm3 Platelet count greater than 100,000/mm3 Hepatic: SGOT and SGPT no greater than 2 times upper limit of normal Alkaline phosphatase no greater than 2 times upper limit of normal Bilirubin no greater than 2 mg/dL Renal: Creatinine no greater than 2.5 mg/dL Other: No known hypersensitivity to porphyrins Not pregnant Fertile patients must use effective birth control

PRIOR CONCURRENT THERAPY: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1995-02; Primary Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley L. Hicks, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States